CLINICAL TRIAL: NCT01570205
Title: The Safety, Tolerability and Pharmacokinetics of a Single Intravenous Infusion of 10, 40, and 80 µg/kg XG-102 Administered to Healthy Male Volunteers in a Randomized, Double Blind, Placebo Controlled, Dose Escalating Phase I Study
Brief Title: Safety, Tolerability and PK of a Single iv Infusion of 10, 40, and 80 µg/kg XG-102 Administered to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xigen SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDD-1002-024
Record Dates: First submitted 2012-03-29; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — D-JNKI-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- XG-102 10 µg/kg (Experimental)
  Interventions: Drug: XG-102
- XG-102 40 µg/kg (Experimental)
  Interventions: Drug: XG-102
- XG-102 80 µg/kg (Experimental)
  Interventions: Drug: XG-102
- placebo (Placebo Comparator)
  Interventions: Drug: XG-102

INTERVENTIONS:
Drug: XG-102 — single intravenous infusion

SUMMARY:
The objective of the study is to investigate safety, tolerability, and pharmacokinetics of XG-102 following iv infusion of single escalating dose of 10, 40, and 80 µg/kg XG-102 to healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age ≥ 18 to ≤ 45 years
* BP: 100 - 150 mm Hg systolic, 50 - 95 mm Hg diastolic and pulse rate: 50 - 100 bpm.
* Body mass index between 18.5 and 30.0 kg/m2 and body weight in the 50 - 100 kg range.
* Are able to communicate and co-operate with the Investigator and his/her staff
* Healthy on the basis of medical history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12 lead ECG readings
* Written informed consent obtained
* Male subjects with partners of childbearing potential have to use adequate contraception during, and for at least the four weeks after administration of study medication.

Exclusion Criteria:

* Heavy smokers, i.e. more than 10 cigarettes per day
* Participation in a clinical trial during the previous 4 weeks
* Loss of 500 mL blood or more during the 3 month period before the screening visit of the study
* Existence of any surgical or medical condition which might relevantly interfere with the subject safety, the distribution, metabolism or excretion of the drug or the study assessments, i.e. impaired renal or hepatic function, diabetes mellitus, thyroid function abnormalities including abnormal thyroid hormone values in the Screening evaluation, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
* History of alcohol or drug abuse in the last 3 years.
* Positive results of the drug Screening.
* Clinically significant abnormal laboratory values at the Screening or baseline evaluation.
* A history of any serious adverse reaction or hypersensitivity to any drug or other medicines
* Presence or history of any allergy requiring acute or chronic treatment (seasonal allergic rhinitis which requires no treatment may be tolerated).
* Positive results from serology examination for HBV, HCV, HIV or tuberculosis
* History of serious mental disorders.
* Need of any prescription medication within 30 days prior to the administration of the drug and/or nonprescription medication within 7 days prior to the administration of the drug or anticipated need for any concomitant medication during the study.
* Volunteers who are unwilling to comply with the provisions of this protocol
* Symptoms of a significant (upon Investigator's medical judgment) somatic or mental illness in the two week period preceding drug administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety of XG-102 | 1 month
  Safety of XG-102 assessed by incidence and intensity of adverse events, clinical laboratory evaluations, vital signs, ECG, phaysical examination, ocular examination

SECONDARY OUTCOMES:
Pharmacokinetics | 16 time-points up to 24 hours
  Pharmacokinetic profile will be evaluated by determination of Cmax, AUC, Half-life, Clearance , Volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — Covance Clinical Research
Locations (1):
- Covance Clinical Research, Allschwil, Canton of Basel-City, Switzerland